CLINICAL TRIAL: NCT02408055
Title: A Phase I Study to Assess the Mass Balance Recovery, Pharmacokinetics, Metabolism and Excretion of 14C-TA-8995 in Healthy Male Subjects
Brief Title: ADME Study in Healthy Male Subjects With TA-8995
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Xention Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TA-8995-07
Record Dates: First submitted 2015-02-25; First posted 2015-04-03 (Estimated); Last update posted 2016-10-03 (Estimated); Status verified 2016-09

CONDITIONS: Dyslipidemia
MeSH Terms: conditions — Dyslipidemias | interventions — TA-8995

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Radiolabelled TA-8995 (Experimental)
  Interventions: Drug: TA-8995

INTERVENTIONS:
Drug: TA-8995

SUMMARY:
A study to measure the absorption, metabolism and excretion of a single dose of radiolabelled TA-8995 (10mg) in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects

Exclusion Criteria:

* Clinically significant abnormalities

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-06; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
AUC of TA-8995 | 35 days
Mass balance recovery of total radioactivity from excreta for radiolabelled TA-8995 | 35 days
Measure the amount of radiolabelled TA-8995 recovered from urine and faeces. | 35 days
Measure the levels of major metabolites of TA-8995 in plasma, urine and faeces after oral administration of radiolabelled TA-8995 | 35 days
Elimination of half-life of radiolabelled TA-8995 | 35 days

SECONDARY OUTCOMES:
Number of adverse events | 35 days

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Brooks, Principal Investigator — Covance
Locations (1):
- Covance Clinical Research Unit Ltd, Leeds, United Kingdom